CLINICAL TRIAL: NCT01644630
Title: A Randomized Controlled Clinical Trial Comparing Cemented Versus Screw-retained Implant-supported Single Crowns With Customized Zirconia Abutments
Brief Title: To Compare Cemented Versus Screw-retained Implant-supported Single Crowns With Customized Zirconia Abutments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-0147
Record Dates: First submitted 2012-07-09; First posted 2012-07-19 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Implant-supported Single Crowns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cemented single crowns (Active Comparator): Cemented single crown: zirconia abutment (Straumann Cares abutment) with an all-ceramic lithium disilicate crown
  Interventions: Procedure: Cemented crowns
- Screw-retained single crown (Active Comparator): Screw-retained single crown: zirconia abutment (Straumann Cares abutment), directly veneered with veneering ceramic
  Interventions: Procedure: Screw-retained crowns

INTERVENTIONS:
Procedure: Cemented crowns — The final lithium disilicate crowns will be cemented with an adhesive cement after tightening the abutments with the torque indicated by the manufacturer and closing the screw access hole with white guttapercha. The abutment will be cleaned with ethanol. A retraction cord will be placed for cementation if indicated. The crown will be etched with hydrofluoric acid and subsequently silanized. A sufficient amount of cement will be filled in the crown without creating major excesses. When the crown is seated correctly, the cement will be light-cured for a few seconds to facilitate the removal of the now hard excess cement.
  - Excess cement will be meticulously removed with a carbon scaler. The removal of all excess cement will be checked with an X-ray and by visual and tactile inspection.
  Arms: Cemented single crowns
Procedure: Screw-retained crowns — The screw-retained crowns will be inserted and tightened with the torque indicated by the manufacturer. The screw access hole will to be closed with white guttapercha and a composite filling (Filtek, 3M ESPE).
  Arms: Screw-retained single crown

SUMMARY:
The aim of this study is to test whether or not the use of screw-retained implant crowns on customized zirconia abutments results in biological, technical and esthetic outcomes similar to those obtained with cemented all-ceramic crowns on customized zirconia abutments, both made with a computer-aided design and manufacturing procedure (CAD/CAM).

The null-hypotheses is that marginal bone level change is equal at screw-retained and cemented crowns

ELIGIBILITY:
Inclusion Criteria:

* Single-tooth Straumann Bone Level in the anterior maxilla or mandible
* At least one adjacent natural tooth present
* Implant position enabling both screw-retained and cemented crown
* Informed consent signed

Exclusion Criteria:

* Smoking more than 15 cigarettes a day
* Poor oral hygiene (Plaque index over 30%)
* Pregnancy at the date of inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-07-27 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Marginal bone level | 5 years
  The bone level represents an indicator of the osseointegration and biological success of the implant.

SECONDARY OUTCOMES:
Biological, technical and esthetic outcome | up to 5 years
  Radiographic bone level after 1 and 3 years
Biological, technical and esthetic outcome | up to 5 years
  implant survival after 1, 3 and 5 years
Biological, technical and esthetic outcome | up to 5 years
  rate of biological complications after 1, 3 and 5 years
Biological, technical and esthetic outcome | up to 5 years
  rate of technical complications after 1, 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Thoma, Prof. Dr., Principal Investigator — Clinic of Reconstructive Dentistry
Locations (1):
- Clinic of Reconstructive Dentistry, Zurich, Switzerland